CLINICAL TRIAL: NCT03066024
Title: Electroencephalogram Dynamics in Children During Different Levels of Anesthetic Depth
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Hospital director of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: Retro-Child
Record Dates: First submitted 2017-02-10; First posted 2017-02-28 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Depth of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents: Children and adolescents for elective surgery

SUMMARY:
As part of the clinical routine of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM in the Charité - University Medicine Berlin intraoperative electroencephalography data and clinical routine data are recorded and evaluated in surgical children and adolescents according to different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents undergoing surgery procedure

Exclusion Criteria:

* Neurosurgery
* Pre-existing neurological conditions

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents during anaesthesia / surgery procedure
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Electroencephalography monitoring changes | Up to the end of surgery

SECONDARY OUTCOMES:
Anesthetic depth | Up to the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Belrin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No